CLINICAL TRIAL: NCT00658021
Title: Safety and Efficacy of Exenatide as Monotherapy and Adjunctive Therapy to Oral Antidiabetic Agents in Adolescents With Type 2 Diabetes.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D5550C00002; H8O-MC-GWBQ (Other: company identifier)
Record Dates: First submitted 2008-04-08; First posted 2008-04-14 (Estimated); Results first posted 2020-12-01 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-10

CONDITIONS: Type 2 Diabetes
Keywords: diabetes; adolescents; exenatide; Astra Zeneca
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Subcutaneous injection, twice a day
  Interventions: Drug: Placebo
- Exenatide 5 µg (Experimental): Subcutaneous injection, twice a day
  Interventions: Drug: Exenatide
- Exenatide 10 µg (Experimental): Subcutaneous injection, twice a day
  Interventions: Drug: Exenatide

INTERVENTIONS:
Drug: Placebo — Subcutaneous injection, twice a day
  Arms: Placebo
Drug: Exenatide — Subcutaneous injection, 5 µg, twice a day
  Arms: Exenatide 5 µg
Drug: Exenatide — Subcutaneous injection,10 µg, twice a day
  Arms: Exenatide 10 µg

SUMMARY:
The primary objective of this study is to test the hypothesis that glycemic control, as measured by change in hemoglobin A1c (HbA1c) from baseline to endpoint, with exenatide is superior to that of placebo after 28 weeks of treatment in adolescent patients with type 2 diabetes who are naïve to antidiabetes agents, or patients who are being treated with metformin, an SU, or a combination of metformin and an SU

ELIGIBILITY:
Inclusion Criteria-patients are eligible to be included in the study only if they meet all of the following criteria:

* are a male or a female between ages 10 to 17 years, inclusive. The number of patients ≥17 years of age will be limited to no more than 10% of patients in each treatment arm
* have a history of type 2 diabetes with the original diagnosis based on at least one American Diabetes Association (ADA) diagnostic criteria
* have been treated with metformin, an SU, or both metformin and an SU (with or without diet and exercise), for at least 3 months or are naïve to anti-diabetes agents and being treated with diet and exercise alone. The dose of oral agent(s) should be stable for the 30 days prior to the screening visit
* have fasting C-peptide >0.6 ng/mL
* have HbA1c between 6.5% and 10.5%, inclusive.

Disease Diagnostic Criteria-for the purposes of this study, patients with type 2 diabetes are defined by:

* diagnosis of type 2 diabetes, as determined by ADA diagnostic criteria and antibody testing, documented and confirmed in the patient's medical record, which includes laboratory determinations consistent with one or more of the following in the patient's medical history
* fasting blood glucose 126 mg/dL (7.0 mmol/L)
* random blood glucose 200 mg/dL (11.1 mmol/L)
* two-hour OGTT (Oral Glucose Tolerance Test) ≥ 200 mg/dL (11.1 mmol/L) AND one or more of the following: no antibodies to GAD65 OR no antibodies to islet cell antigen (ICA512).

Exclusion Criteria-patients will be excluded from the study if they meet any of the following criteria:

* have previously been exposed to exenatide or, completed or withdrawn from this study or any other study investigating exenatide
* are unwilling or unable to inject the study medication
* currently use inhaled steroids at a dose equal to or above 1000g Flovent (fluticasone propionate) daily
* have used oral steroids within the last 60 days or more than 20 days use within the past year
* have used any weight loss medication(s) within 30 days of screening
* have used insulin for more than 10 weeks during the 3 months prior to screening
* have history of renal disease, or serum creatinine >1.6 mg/dL (141.4 µmol/L) (males) or >1.4 mg/dL (123.8 µmol/L) (females)
* have hepatic dysfunction, defined by aspartate (AST) or alanine (ALT) transaminase >3.0 times the upper limit of normal (ULN).

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 122 (Actual)
Dates: Start 2008-05-30 (Actual); Primary Completion 2019-04-18 (Actual); Study Completion 2020-04-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (52):
- United States (30):
  - Research Site, Birmingham, Alabama
  - Research Site, Tucson, Arizona
  - Research Site, Los Angeles, California
  - Research Site, Montclair, California
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, Santa Ana, California
  - Research Site, Aurora, Colorado
  - Research Site, Melbourne, Florida
  - Research Site, Miami, Florida
  - Research Site, Miami Lakes, Florida
  - Research Site, Orlando, Florida
  - Research Site, Pensacola, Florida
  - Research Site, Tallahassee, Florida
  - Research Site, Dalton, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Wichita, Kansas
  - Research Site, Dearborn, Michigan
  - Research Site, Kansas City, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Reno, Nevada
  - Research Site, Jamaica, New York
  - Research Site, Greenville, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Memphis, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Spokane, Washington
- Brazil (3):
  - Research Site, Fortaleza
  - Research Site, Juiz de Fora
  - Research Site, Santo André
- India (3):
  - Research Site, Ahmedabad
  - Research Site, Bangalore
  - Research Site, Pune
- Mexico (7):
  - Research Site, Aguascalientes
  - Research Site, Culiacán
  - Research Site, Guadalajara
  - Research Site, Monterrey
  - Research Site, San Juan del Río
  - Research Site, Tamaupilas
  - Research Site, Tampico
- Research Site, Quezon City, Philippines
- Russia (3):
  - Research Site, Moscow
  - Research Site, Tomsk
  - Research Site, Ufa
- South Africa (4):
  - Research Site, Moloto South
  - Research Site, Paarl
  - Research Site, Pretoria
  - Research Site, Verulam
- Research Site, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment.
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Clinical_Study_Protocol_redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5550C00002&attachmentIdentifier=305e146c-5f7f-45a2-85e8-a10dafda43fb&fileName=D5550C00002_CSP_redacted.pdf&versionIdentifier=
- See also: Statistical Analysis Plan_redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5550C00002&attachmentIdentifier=6cfc1d5f-a256-4d8b-8b54-6944c1993205&fileName=D5550C00002_Statistical_Analysis_Plan.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in adolescents (aged 10 to 17 years inclusive) with type 2 diabetes who were naïve to antidiabetics, or were receiving metformin, an sulfonylurea (SU) or a combination of metformin and an SU in 7 countries (Brazil, India, South Korea, Mexico, Russia, the United States and South Africa) between 30 May 2008 and 01 April 2020.
Pre-assignment Details: The study commenced with a 1-week, single-blind, injectable placebo lead-in period before participants were randomized to 1 of 3 treatment groups: exenatide 5 microgram (mcg) twice daily, exenatide 10 mcg twice daily, or placebo twice daily. A total of 122 participants were randomized in this study.
Groups:
- Exenatide 5 mcg: Adolescent participants received exenatide 5 mcg subcutaneous (SC) injection twice daily for 28 weeks. In the Safety Follow-up Period, participants with a height difference of at least 5 millimeter (mm) between Day 1 and Week 28 visits returned for study visits every 6 months for up to 3 years after completion of the treatment period.
- Exenatide 10 mcg: Adolescent participants received exenatide 5 mcg SC injection twice daily for 4 weeks after randomization. At the end of 4 weeks post-randomization, participants received exenatide 10 mcg SC injection twice daily for next 24 weeks. In the Safety Follow-up Period, participants with a height difference of at least 5 mm between Day 1 and Week 28 visits returned for study visits every 6 months for up to 3 years after completion of the treatment period.
- Placebo: Adolescent participants received placebo matching with exenatide 5 mcg or 10 mcg SC injection twice daily for 28 weeks. In the Safety Follow-up Period, participants with a height difference of at least 5 mm between Day 1 and Week 28 visits returned for study visits every 6 months for up to 3 years after completion of the treatment period.
Period: 28-Week Treatment Period
Arm/Group | Exenatide 5 mcg | Exenatide 10 mcg | Placebo
Started (Randomized to treatment.) | 42 | 38 | 42
Received Treatment | 40 | 38 | 42
Completed (Completed the Week 28 treatment period.) | 31 | 25 | 25
Not Completed | 11 | 13 | 17
Not completed — Adverse Event | 3 | 1 | 0
Not completed — Developed study withdrawal criteria | 0 | 2 | 0
Not completed — Protocol Violation | 0 | 2 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 3
Not completed — Physician Decision | 1 | 2 | 1
Not completed — Withdrawal by parent/guardian | 1 | 1 | 1
Not completed — Loss of glucose control | 1 | 1 | 10
Not completed — Other | 2 | 3 | 1
Not completed — Did not receive treatment | 2 | 0 | 0
Period: Long-term Safety Follow-up Period
Arm/Group | Exenatide 5 mcg | Exenatide 10 mcg | Placebo
Started (Entered safety follow-up period.) | 7 (Entered safety follow-up period.) | 5 (Entered safety follow-up period.) | 7 (Entered safety follow-up period.)
Completed (Completed safety follow-up period.) | 7 | 2 | 7
Not Completed | 0 | 3 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Physician Decision | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: The Intent-To-Treat analysis set included all randomized participants.
Groups:
- Exenatide 5 mcg: Adolescent participants received exenatide 5 mcg SC injection twice daily for 28 weeks. In the Safety Follow-up Period, participants with a height difference of at least 5 mm between Day 1 and Week 28 visits returned for study visits every 6 months for up to 3 years after completion of the treatment period.
- Total: Total of all reporting groups
Arm/Group | Exenatide 5 mcg | Exenatide 10 mcg | Placebo | Total
Number analyzed (Participants) | 42 | 38 | 42 | 122
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.7 (1.94) | 14.0 (1.95) | 14.4 (1.82) | 14.0 (1.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 22 | 29 | 82
  Male | 11 | 16 | 13 | 40
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Ethnicity not collected and Hispanic was collected as a Race in this study.
  Participants
    White | 7 | 5 | 13 | 25
    Black or African American | 14 | 8 | 7 | 29
    Asian | 3 | 2 | 5 | 10
    American Indian or Alaska Native | 0 | 1 | 0 | 1
    Hispanic | 18 | 22 | 17 | 57

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Change From Baseline in Glycated Hemoglobin A1c (HbA1c) at Week 28
Description: Change from baseline in HbA1c is reported as adjusted least square (LS) mean values at Week 28. Baseline is defined as the last non-missing assessment (scheduled or unscheduled) on or prior to the first dose of study medication. A mixed model with repeated measures (MMRM) analysis was performed, excluding measurements after initiation of rescue medication and study drug discontinuation.
Time Frame: Baseline (Day 1) and Week 28
Population: The Evaluable Analysis Set included all randomized participants who received at least 1 dose of randomized study medication and had a baseline and at least 1 post-baseline HbA1c assessment. For analysis of efficacy, a decision was made with agreement by the European Medicines Agency and the Food and Drug Administration to pool participants from both exenatide groups (Total EBID) and compare this pooled group with placebo.
Measure: Least Squares Mean (Standard Error); unit: percentage (%HbA1c)
Groups:
- Total Exenatide Twice Daily (EBID): Efficacy data from participants from both exenatide groups (Total EBID) was pooled for comparison with placebo.
  Adolescent participants received exenatide 5 mcg SC injection twice daily for 28 weeks; or Adolescent participants received exenatide 5 mcg SC injection twice daily for 4 weeks after randomization. At the end of 4 weeks post-randomization, participants received exenatide 10 mcg SC injection twice daily for next 24 weeks.
Arm/Group | Total Exenatide Twice Daily (EBID) | Placebo
Number analyzed (Participants) | 78 | 42
percentage (%HbA1c) | 0.11 (0.215) | 0.38 (0.293)
Statistical Analysis 1: Comparison: Total Exenatide Twice Daily (EBID) vs Placebo; Adjusted LS mean and treatment group difference in the change from baseline values at visit are obtained from a MMRM including treatment, baseline HbA1c, background diabetes therapy strata, week of visit, baseline HbA1c-by-visit interaction and treatment-by-visit interaction as fixed effects using an unstructured covariance matrix; Test type: Superiority; p = 0.444, Mixed Models Analysis; LS Mean Difference = -0.28, 95% CI 2-sided [-1.01 to 0.45], Standard Error of Mean 0.363

2. Primary Outcome: Number of Participants With Post-Treatment Adverse Events of Special Interest (AESI) During Safety Follow-up Period
Description: Post-treatment adverse events (AEs) were defined as AEs that started or worsened during the off-treatment period (Safety Follow-up Period), which was defined as the day after the Week 28/early discontinuation (ED) visit to the date of completion of the Safety Follow-up Period. The AESIs recorded were as follows: hematological malignancies, thyroid neoplasms, pancreas neoplasms, aplastic anemia, pancreatitis, pregnancy and pregnancy outcomes (including congenital anomalies).
Time Frame: From 1 day after the Week 28/ED visit to 3 years after Week 28/ED visit.
Population: The Safety Follow-up Analysis Set included all participants who had at least 1 safety follow-up period assessment visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Exenatide 5 mcg | Exenatide 10 mcg | Placebo
Number analyzed (Participants) | 7 | 5 | 7
Participants | 0 | 0 | 0

3. Secondary Outcome: Percentage of Participants Achieving HbA1c Goals of < 7%, <= 6.5%, and < 6.5% Through Week 28
Description: The percentage of participants achieving HbA1c goals of < 7%, <= 6.5%, and < 6.5% through Week 28 were compared between treatments using the Cochran-Mantel-Haenszel (CMH) procedure, in which screening HbA1c strata and background diabetes therapy strata served as the stratification factors. The CMH analysis excluded measurements after initiation of rescue medication and study drug discontinuation with missing data treated as non-responder.
Time Frame: Weeks 0, 4, 12, 20 and 28
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Total Exenatide Twice Daily (EBID) | Placebo
Number analyzed (Participants) | 78 | 42
percentage of participants
  HbA1c < 7%: Week 0 | 37.2 [26.5 to 47.9] | 38.1 [23.4 to 52.8]
  HbA1c < 7%: Week 4 | 44.9 [33.8 to 55.9] | 42.9 [27.9 to 57.8]
  HbA1c < 7%: Week 12 | 43.6 [32.6 to 54.6] | 33.3 [19.1 to 47.6]
  HbA1c < 7%: Week 20 | 35.9 [25.3 to 46.5] | 35.7 [21.2 to 50.2]
  HbA1c < 7%: Week 28 | 33.3 [22.9 to 43.8] | 28.6 [14.9 to 42.2]
  HbA1c <=6.5%: Week 0 | 17.9 [9.4 to 26.5] | 16.7 [5.4 to 27.9]
  HbA1c <=6.5%: Week 4 | 29.5 [19.4 to 39.6] | 23.8 [10.9 to 36.7]
  HbA1c <=6.5%: Week 12 | 33.3 [22.9 to 43.8] | 23.8 [10.9 to 36.7]
  HbA1c <=6.5%: Week 20 | 24.4 [14.8 to 33.9] | 19.0 [7.2 to 30.9]
  HbA1c <=6.5%: Week 28 | 23.1 [13.7 to 32.4] | 19.0 [7.2 to 30.9]
  HbA1c <6.5%: Week 0 | 15.4 [7.4 to 23.4] | 7.1 [0.0 to 14.9]
  HbA1c <6.5%: Week 4 | 26.9 [17.1 to 36.8] | 21.4 [9.0 to 33.8]
  HbA1c <6.5%: Week 12 | 30.8 [20.5 to 41.0] | 19.0 [7.2 to 30.9]
  HbA1c <6.5%: Week 20 | 21.8 [12.6 to 31.0] | 19.0 [7.2 to 30.9]
  HbA1c <6.5%: Week 28 | 23.1 [13.7 to 32.4] | 14.3 [3.7 to 24.9]
Statistical Analysis 1: Comparison: Total Exenatide Twice Daily (EBID) vs Placebo; Treatment difference in HbA1c < 7% at Week 28: Treatment group comparison is based on CMH test stratified by screening HbA1c and background diabetes therapy strata. P-value is from the general association statistics; Test type: Superiority; p = 0.562, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Total Exenatide Twice Daily (EBID) vs Placebo; Treatment difference in HbA1c <= 6.5% at Week 28: Treatment group comparison is based on CMH test stratified by screening HbA1c and background diabetes therapy strata. P-value is from the general association statistics; Test type: Superiority; p = 0.621, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Total Exenatide Twice Daily (EBID) vs Placebo; Treatment difference in HbA1c < 6.5% at Week 28: Treatment group comparison is based on CMH test stratified by screening HbA1c and background diabetes therapy strata. P-value is from the general association statistics; Test type: Superiority; p = 0.229, Cochran-Mantel-Haenszel

4. Secondary Outcome: Adjusted Change From Baseline in Body Weight Through Week 28
Description: Change from baseline in body weight is reported as adjusted LS mean values at Weeks 4, 12, 20 and 28. Baseline is defined as the last non-missing assessment (scheduled or unscheduled) on or prior to the first dose of study medication. A MMRM analysis was performed, excluding measurements after initiation of rescue medication and study drug discontinuation.
Time Frame: Baseline (Day 1) up to Week 28
Population: The Full Analysis Set included all randomized participants who received at least 1 dose of randomized study medication. For analysis of efficacy, a decision was made with agreement by the European Medicines Agency and the Food and Drug Administration to pool participants from both exenatide groups (Total EBID) and compare this pooled group with placebo.
Measure: Least Squares Mean (Standard Error); unit: kilogram
Arm/Group | Total Exenatide Twice Daily (EBID) | Placebo
Number analyzed (Participants) | 78 | 42
kilogram
  Week 4 | -0.89 (0.196) | 0.04 (0.260)
  Week 12 | -1.09 (0.401) | -0.42 (0.534)
  Week 20 | -0.71 (0.559) | -0.33 (0.755)
  Week 28 | -0.81 (0.632) | -0.36 (0.857)
Statistical Analysis 1: Comparison: Total Exenatide Twice Daily (EBID) vs Placebo; Treatment difference in body weight at Week 4: Adjusted LS mean and treatment group difference in the change from baseline values at visit are obtained from a MMRM including treatment, baseline body weight, screening HbA1c strata, background diabetes therapy strata, week of visit, baseline body weight-by visit interaction and treatment-by-visit interaction as fixed effects using an unstructured covariance matrix; Test type: Superiority; p = 0.005, Mixed Models Analysis; LS Mean Difference = -0.93, 95% CI 2-sided [-1.58 to -0.28], Standard Error of Mean 0.327
Statistical Analysis 2: Comparison: Total Exenatide Twice Daily (EBID) vs Placebo; Treatment difference in body weight at Week 12: Adjusted LS mean and treatment group difference in the change from baseline values at visit are obtained from a MMRM including treatment, baseline body weight, screening HbA1c strata, background diabetes therapy strata, week of visit, baseline body weight-by visit interaction and treatment-by-visit interaction as fixed effects using an unstructured covariance matrix; Test type: Superiority; p = 0.314, Mixed Models Analysis; LS Mean Difference = -0.68, 95% CI 2-sided [-2.00 to 0.65], Standard Error of Mean 0.669
Statistical Analysis 3: Comparison: Total Exenatide Twice Daily (EBID) vs Placebo; Treatment difference in body weight at Week 20: Adjusted LS mean and treatment group difference in the change from baseline values at visit are obtained from a MMRM including treatment, baseline body weight, screening HbA1c strata, background diabetes therapy strata, week of visit, baseline body weight-by visit interaction and treatment-by-visit interaction as fixed effects using an unstructured covariance matrix; Test type: Superiority; p = 0.692, Mixed Models Analysis; LS Mean Difference = -0.37, 95% CI 2-sided [-2.24 to 1.50], Standard Error of Mean 0.940
Statistical Analysis 4: Comparison: Total Exenatide Twice Daily (EBID) vs Placebo; Treatment difference in body weight at Week 28: Adjusted LS mean and treatment group difference in the change from baseline values at visit are obtained from a MMRM including treatment, baseline body weight, screening HbA1c strata, background diabetes therapy strata, week of visit, baseline body weight-by visit interaction and treatment-by-visit interaction as fixed effects using an unstructured covariance matrix; Test type: Superiority; p = 0.679, Mixed Models Analysis; LS Mean Difference = -0.44, 95% CI 2-sided [-2.56 to 1.68], Standard Error of Mean 1.065

5. Secondary Outcome: Adjusted Change From Baseline in Fasting Serum Glucose (FSG) at Week 28
Description: Change from baseline in FSG is reported as adjusted LS mean values at Week 28. Baseline is defined as the last non-missing assessment (scheduled or unscheduled) on or prior to the first dose of study medication. An analysis of covariance (ANCOVA) analysis was performed, excluding measurements after initiation of rescue medication and study drug discontinuation.
Time Frame: Baseline (Day 1) and Week 28
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: millimoles per liter (mmol/L)
Arm/Group | Total Exenatide Twice Daily (EBID) | Placebo
Number analyzed (Participants) | 78 | 42
millimoles per liter (mmol/L) | 0.791 (0.4010) | 1.072 (0.5466)
Statistical Analysis 1: Comparison: Total Exenatide Twice Daily (EBID) vs Placebo; Adjusted LS Mean and treatment group difference in the change from baseline values at Week 28 are obtained from multiple imputation ANCOVA including treatment, baseline fasting serum glucose, screening HbA1c strata and background diabetes therapy strata as fixed effects; Test type: Superiority; p = 0.679, ANCOVA; LS Mean Difference = -0.281, 95% CI 2-sided [-1.614 to 1.052], Standard Error of Mean 0.6800

6. Secondary Outcome: Adjusted Change From Baseline in Self-Monitored Blood Glucose (SMBG) at Week 28
Description: Change from baseline in SMBG measurements are reported as adjusted LS mean values at Week 28. SMBG measurements were taken before (pre-prandial) and 2 hours after (post-prandial) the 2 main meals of the day on 3 separate days during the week before baseline (Day 1) and Week 28. Post-prandial excursions were calculated as the difference between the pre-prandial and post-prandial blood glucose concentrations (post-prandial - pre-prandial) and averaged (mean) over the 2 main meals over the 3 separate days in each period. Baseline is defined as the last non-missing assessment (scheduled or unscheduled) on or prior to the first dose of study medication. An ANCOVA analysis was performed, excluding measurements after initiation of rescue medication and study drug discontinuation.
Time Frame: Pre-meal and 2 hours post-meal on Baseline (Day 1) and Week 28
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Total Exenatide Twice Daily (EBID) | Placebo
Number analyzed (Participants) | 78 | 42
mmol/L
  Pre-meal SMBG | -0.699 (0.2709) | -0.888 (0.4511)
  Post-meal SMBG | -1.029 (0.2722) | -1.542 (0.4503)
  Post-prandial excursion SMBG | -0.181 (0.2107) | -0.391 (0.3418)
  Overall SMBG | -0.877 (0.2468) | -1.193 (0.4117)
Statistical Analysis 1: Comparison: Total Exenatide Twice Daily (EBID) vs Placebo; Treatment difference for pre-meal SMBG: Adjusted LS Mean and treatment group difference in the change from baseline values at Week 28 are obtained from multiple imputation ANCOVA including treatment, baseline SMBG measure, screening HbA1c strata and background diabetes therapy strata as fixed effects; Test type: Superiority; p = 0.714, ANCOVA; LS Mean Difference = 0.189, 95% CI 2-sided [-0.821 to 1.199], Standard Error of Mean 0.5151
Statistical Analysis 2: Comparison: Total Exenatide Twice Daily (EBID) vs Placebo; Treatment difference for post-meal SMBG: Adjusted LS Mean and treatment group difference in the change from baseline values at Week 28 are obtained from multiple imputation ANCOVA including treatment, baseline SMBG measure, screening HbA1c strata and background diabetes therapy strata as fixed effects; Test type: Superiority; p = 0.329, ANCOVA; LS Mean Difference = 0.513, 95% CI 2-sided [-0.516 to 1.541], Standard Error of Mean 0.5245
Statistical Analysis 3: Comparison: Total Exenatide Twice Daily (EBID) vs Placebo; Treatment difference for post-prandial excursion SMBG: Adjusted LS Mean and treatment group difference in the change from baseline values at Week 28 are obtained from multiple imputation ANCOVA including treatment, baseline SMBG measure, screening HbA1c strata and background diabetes therapy strata as fixed effects; Test type: Superiority; p = 0.601, ANCOVA; LS Mean Difference = 0.210, 95% CI 2-sided [-0.577 to 0.997], Standard Error of Mean 0.4015
Statistical Analysis 4: Comparison: Total Exenatide Twice Daily (EBID) vs Placebo; Treatment difference for overall SMBG: Adjusted LS Mean and treatment group difference in the change from baseline values at Week 28 are obtained from multiple imputation ANCOVA including treatment, baseline SMBG measure, screening HbA1c strata and background diabetes therapy strata as fixed effects; Test type: Superiority; p = 0.505, ANCOVA; LS Mean Difference = 0.316, 95% CI 2-sided [-0.615 to 1.248], Standard Error of Mean 0.4749

7. Secondary Outcome: Adjusted Change From Baseline in Fasting Serum Insulin at Week 28
Description: Change from baseline in fasting serum insulin is reported as adjusted LS mean values at Week 28. Baseline is defined as the last non-missing assessment (scheduled or unscheduled) on or prior to the first dose of study medication. An ANCOVA analysis was performed, excluding measurements after initiation of rescue medication and study drug discontinuation.
Time Frame: Baseline (Day 1) and Week 28
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: picomoles per liter
Arm/Group | Total Exenatide Twice Daily (EBID) | Placebo
Number analyzed (Participants) | 78 | 42
picomoles per liter | 1.67 (25.323) | 12.49 (34.825)
Statistical Analysis 1: Comparison: Total Exenatide Twice Daily (EBID) vs Placebo; Adjusted LS Mean and treatment group difference in the change from baseline values at Week 28 are obtained from multiple imputation ANCOVA including treatment, baseline fasting serum insulin, screening HbA1c strata and background diabetes therapy strata as fixed effects; Test type: Superiority; p = 0.802, ANCOVA; LS Mean Difference = -10.82, 95% CI 2-sided [-95.48 to 73.84], Standard Error of Mean 43.187

8. Secondary Outcome: Adjusted Change From Baseline in Homeostasis Model Assessments - Beta-Cell Function (HOMA-B) and Insulin Sensitivity (HOMA-S) at Week 28
Description: Change from baseline in HOMA-B and HOMA-S are reported as adjusted LS mean values at Week 28. Baseline is defined as the last non-missing assessment (scheduled or unscheduled) on or prior to the first dose of study medication. An ANCOVA analysis was performed, excluding measurements after initiation of rescue medication and study drug discontinuation.
Time Frame: Baseline (Day 1) and Week 28
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: percentage (%HOMA-B and %HOMA-S)
Arm/Group | Total Exenatide Twice Daily (EBID) | Placebo
Number analyzed (Participants) | 78 | 42
percentage (%HOMA-B and %HOMA-S)
  HOMA-B | -25.93 (10.404) | -22.10 (14.885)
  HOMA-S | -3.18 (2.172) | -2.90 (3.117)
Statistical Analysis 1: Comparison: Total Exenatide Twice Daily (EBID) vs Placebo; Treatment difference for HOMA-B: Adjusted LS Mean and treatment group difference in the change from baseline values at Week 28 are obtained from multiple imputation ANCOVA including treatment, baseline %HOMA-B, screening HbA1c strata and background diabetes therapy strata as fixed effects; Test type: Superiority; p = 0.836, ANCOVA; LS Mean Difference = -3.84, 95% CI 2-sided [-40.19 to 32.51], Standard Error of Mean 18.542
Statistical Analysis 2: Comparison: Total Exenatide Twice Daily (EBID) vs Placebo; Treatment difference for HOMA-S: Adjusted LS Mean and treatment group difference in the change from baseline values at Week 28 are obtained from multiple imputation ANCOVA including treatment, baseline %HOMA-S, screening HbA1c strata and background diabetes therapy strata as fixed effects; Test type: Superiority; p = 0.941, ANCOVA; LS Mean Difference = -0.28, 95% CI 2-sided [-7.82 to 7.26], Standard Error of Mean 3.846

9. Secondary Outcome: Percentage of Participants Discontinuing the Study Due to Failure to Maintain Glycemic Control Through Week 28
Description: Participants were discontinued from the study due to failure to maintain glycemic control if either discontinuation reason on summary case report form was "Loss of glucose control" or AE with lower level Medical Dictionary for Regulatory Activities (MedDRA) term "Loss of control of blood sugar" or "Hyperglycaemia" leading to study drug discontinuation, using MedDRA Version 23.0.
Time Frame: Weeks 2, 4, 8, 12, 16, 20, 24 and 28
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Total Exenatide Twice Daily (EBID) | Placebo
Number analyzed (Participants) | 78 | 42
percentage of participants
  Week 2 | 0 | 0
  Week 4 | 0 | 2.4
  Week 8: number analyzed (Participants) | 78 | 41
  Week 8 | 0 | 0
  Week 12: number analyzed (Participants) | 78 | 40
  Week 12 | 1.4 | 5.0
  Week 16: number analyzed (Participants) | 78 | 36
  Week 16 | 1.4 | 0
  Week 20: number analyzed (Participants) | 78 | 34
  Week 20 | 0 | 14.7
  Week 24: number analyzed (Participants) | 78 | 29
  Week 24 | 0 | 6.9
  Week 28: number analyzed (Participants) | 78 | 26
  Week 28 | 1.6 | 0

ADVERSE EVENTS:
Time Frame: Serious AEs: From first dose of study drug (Day 1) up to 30 days after last dose of study drug, approximately 32 weeks. Non-serious AEs: From first dose of study drug (Day 1) up to 1 day after last dose of study drug, approximately 28 weeks.
Description: The Safety Analysis Set included all participants who received at least 1 dose of randomized study medication.
  Treatment-emergent AEs (TEAEs) are reported. A TEAE was defined as an AE starting (or worsening) after the first dose of randomized study medication through the end of treatment + 1 day for non-serious AEs or + 30 days for serious AEs.
Groups:
- Exenatide 5 mcg: Adolescent participants received exenatide 5 mcg SC injection twice daily for 28 weeks.
- Exenatide 10 mcg: Adolescent participants received exenatide 5 mcg SC injection twice daily for 4 weeks after randomization. At the end of 4 weeks post-randomization, participants received exenatide 10 mcg SC injection twice daily for next 24 weeks.
- Placebo: Adolescent participants received placebo matching with exenatide 5 mcg or 10 mcg SC injection twice daily for 28 weeks.
Arm/Group | Exenatide 5 mcg | Exenatide 10 mcg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/37 | 0/42
Serious Adverse Events (participants affected / at risk) | 3/41 | 1/37 | 1/42
Other Adverse Events (participants affected / at risk) | 26/41 | 24/37 | 23/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exenatide 5 mcg (N=41) | Exenatide 10 mcg (N=37) | Placebo (N=42)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
Intentional self-injury (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exenatide 5 mcg (N=41) | Exenatide 10 mcg (N=37) | Placebo (N=42)
Ear pain (Ear and labyrinth disorders) | 2 (2) | 2 (2) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 2 (5) | 2 (4)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 3 (3) | 5 (9)
Nausea (Gastrointestinal disorders) | 4 (4) | 11 (15) | 7 (10)
Vomiting (Gastrointestinal disorders) | 2 (2) | 8 (10) | 3 (3)
Pyrexia (General disorders) | 2 (2) | 1 (1) | 3 (3)
Furuncle (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Influenza (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 8 (10) | 2 (4) | 3 (3)
Pharyngitis (Infections and infestations) | 4 (6) | 2 (5) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 4 (4) | 1 (1) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 5 (8) | 3 (3) | 5 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (4) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 2 (3) | 2 (2)
Headache (Nervous system disorders) | 9 (14) | 9 (15) | 11 (27)
Dysmenorrhoea (Reproductive system and breast disorders) | 2 (3) | 3 (4) | 4 (6)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-10-13): https://cdn.clinicaltrials.gov/large-docs/21/NCT00658021/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-22): https://cdn.clinicaltrials.gov/large-docs/21/NCT00658021/SAP_001.pdf